CLINICAL TRIAL: NCT04025359
Title: The Effects of Dronabinol in Opioid-Related Outcomes
Brief Title: Effects of Dronabinol in Opioid Maintained Patients
Acronym: THC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2000027065
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled cross-over human laboratory study. Participants will be asked to come to the testing site for a total of four times: one initial screening session (~ 3 hours) and three test days (~ 6 hours each) where study medication will be administered, separated by at least 72 hours to limit carryover effects for dronabinol administration.
Who Masked: Participant, Investigator
Masking Description: The study medication will be prepared by research pharmacy using over-encapsulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dronabinol 2.5mg (Active Comparator): Dronabinol 2.5mg
  Interventions: Drug: Dronabinol
- Dronabinol 5mg (Active Comparator): Dronabinol 5mg
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol 2.5 mg
  Other Names: Marinol
  Arms: Dronabinol 2.5mg
Drug: Dronabinol — Dronabinol 5 mg
  Other Names: Marinol
  Arms: Dronabinol 5mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Twenty male and female (ages 18-70) participants with OUD currently receiving methadone or buprenorphine will be enrolled. Prior to their daily methadone or buprenorphine dose and thus at trough plasma levels of opioid, participants will receive dronabinol (2.5 mg, 5mg) or placebo. Subsequently, all participants will undergo laboratory testing of opioid-related outcomes. Pain sensitivity will be measured using a technique called the (QST) quantitative sensory testing, which involves the administering heat or cold stimulation. A Short-Form McGill Pain Questionnaire (SF-MPQ) and a pain Visual Analog Scale (VAS). Attentional bias will be measured using a visual probe task. Negative affect will be measured using the Positive and Negative Affect Schedule (PANAS). Cognitive performance will be measured by a comprehensive cognitive battery. The order of study medication administration will be counterbalanced order to minimize carryover effects. On the initial screening day and at the end of medication treatment, blood will be drawn to determine serum cytokine levels. One week after the last study medication dose, a follow-up session will be conducted during which participants will undergo urine toxicology testing and a safety evaluation before final discharge from the study.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled cross-over human laboratory study. Participants will be asked to come to the testing site for a total of four times: one initial screening session (~ 3 hours) and three test days (~ 6 hours each) where study medication will be administered, separated by at least 72 hours to limit carryover effects for dronabinol administration. Twenty male and female participants with OUD on MAT will be asked to arrive at approximately the same time each morning, coordinating with attendance at their opioid maintenance clinic. Subjects will be asked to refrain from using alcoholic beverages and drugs during study participation. Urine screens and breathalyzer measurements will be done before the test sessions to check abstinence from drugs (e.g., cocaine, illicit opioids, benzodiazepines, barbiturates, and amphetamines) and alcohol respectively. Those who are non-compliant will be discharged from the study. To minimize nicotine and withdrawal effects on cognitive performance, subjects who smoke will be advised to continue smoking as usual. Since we will provide a standard breakfast, participants will be asked not to eat for two hour before they arrive for the test sessions. A study nurse will confirm with their respective program that participants did not receive either methadone or buprenorphine that morning, and will call the program when testing is complete to permit dispersal of that day's methadone or buprenorphine dose. On the initial screening day and at the end of medication treatment, blood will be drawn to determine serum cytokine levels. Participants will undergo a variety of cognitive and self-report measures, as well as assessments to confirm restraint from illicit drug use and lack of adverse effects of medication. Prior to their daily methadone or buprenorphine dose and thus at trough plasma levels of opioid, participants will receive dronabinol (10 mg, 20 mg) or placebo. Subsequently, all participants will undergo laboratory testing of measures relevant to vulnerability to relapse, including physiological, subjective and cognitive outcomes. The order of study medication administration will be counterbalanced order to minimize the impact of potential carryover effects between the sessions. To date: 27 subjects completed the approve protocol.

This study was amended to reduce the study drug (dronabinol) to 2.5mg, 5mg, or placebo. This study is active with recruitment continuing under the new doses.

ELIGIBILITY:
Inclusion Criteria:

* Prior exposure to THC or cannabis at least once in the last 10 years; 1-10 times in the last 20 years; or more than 20 times in their lifetime.
* Males and females, Veterans and non-Veterans, aged between 18 and 70.
* Diagnosed with OUD and currently enrolled in methadone or buprenorphine maintenance treatment.
* Capable of providing informed consent in English.
* Compliant in opioid maintenance treatment and on a stable dose for two weeks or longer.
* Not meeting DSM-5 criteria for substance use disorders other than OUD or tobacco use disorder within the last 12 months.
* No current medical problems deemed contraindicated for participation by principal investigator.
* For women, not pregnant as determined by pregnancy screening; not breast-feeding; using acceptable birth control methods.

Exclusion Criteria:

* Currently meeting DSM-5 criteria for cannabis use disorder (CUD).
* History of primary psychotic disorders or other current major psychiatric disorders deemed clinically unstable by the principal investigator.
* Serious medical or neurological illness or treatment for a medical disorder that could interfere with study participation as determined by principal investigator.
* Inability to complete neuropsychological tests.
* A physician will carefully evaluate participants for use of over-the-counter or prescription psychoactive drugs known to affect pain threshold or pain tolerance (including NSAIDS, serotonin-norepinephrine reuptake inhibitors (SNRIs), (e.g. venlafaxine, duloxetine), tricyclic antidepressants (e.g., nortriptyline, amitriptyline), anticonvulsant medications (e.g., topiramate, tegretol), benzodiazepines (e.g., alprazolam, diazepam), and other opioid drugs). Only subjects who are on stable doses of these medications, and whose dosing schedules allow participation in the study visits, will be enrolled. If possible, the morning dose will be administered after the study visit.
* Liver function tests (ALT or AST) greater than 3x normal.
* Contraindications for exposure to cold temperatures, such as Raynaud's phenomenon and hypertension.
* Allergy or serious adverse reaction to cannabis, dronabinol or other cannabinoids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain sensitivity, measured by the Cold Pressor Test (CPT). | up to 6 hours
  Pain threshold and pain tolerance, in seconds.
Pain sensitivity, measured by the Short form of the McGill Pain Questionnaire (SF-MPQ). | up to 6 hours
  Subjective pain measured by the SF-MPQ. The SF-MPQ values range from 0 to 45, with higher values indicating greater pain sensitivity.

SECONDARY OUTCOMES:
Abuse potential, measured by the Drug Effects Questionnaire (DEQ). | up to 6 hours
  The DEQ values range from 0-100, with higher values indicating more prominent subjective drug effects.
Cognitive Performance, measured by the Continuous Performance Test (CPT) | up to 6 hours
  Sustained attention and verbal learning measured by the CPT. The outcome for the CPT is the percent of correct responses, with a higher percentage indicating greater attention and working memory performance.
Cognitive Performance, measured by the Hopkins Verbal Learning Test (HVLT). | up to 6 hours
  Sustained attention and verbal learning measured by the HVLT. The outcome for the HVLT is the immediate total recall, ranging from 0-36, with higher values indicating greater verbal learning.

CONTACTS AND LOCATIONS:
Overall Officials: Joao De Aquino, M.D., Principal Investigator — VA healthcare System West Haven CT
Locations (1):
- VA Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided